CLINICAL TRIAL: NCT06504680
Title: Results of 8 Strand Repair of Flexor Tendon Injuries Zone II With and Without Splinting of the Wrist A Randomized Controlled Trial
Brief Title: Results of 8 Strand Repair of Flexor Tendon Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud Mohamed Abdelrahim, Dr/yasser farouq, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cut flexor zone ll
Record Dates: First submitted 2024-04-03; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Cut Flexor Zone ll Using 8-strand

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splinted cases (Active Comparator): Repair cut flexor zone ll using 8-strand with splint the wrist
  Interventions: Procedure: Repair of flexor tendon injury zone ll using 8- strand
- Non splinting cases (Active Comparator): Repair cut flexor zone ll using 8-strand without splint the wrist
  Interventions: Procedure: Repair of flexor tendon injury zone ll using 8- strand

INTERVENTIONS:
Procedure: Repair of flexor tendon injury zone ll using 8- strand — Repair cut flexor zone ll using 8-strand with and without splinting the wrist

SUMMARY:
Functional results of 8 strand repair of flexor tendon injuries zone II with and without splinting of the wrist

DETAILED DESCRIPTION:
Flexor tendon injuries of the hand, account for 30% of all hand injuries, but are difficult to treat and are associated with frequent poor outcomes . While major progress has been made with the treatment of these injuries, current surgical treatment relies mostly on conventional suturing techniques with variable results, concluding in re-operation rates of 12%, and complication rate of up to 20% Restoration of tendon gliding is the goal when repairing flexor tendon injuries. The tendon forces experienced during postoperative, active flexion exercises are significantly larger than the tendon forces experienced by patients engaging in only passive flexion. Multistrand sutures (typically four- or six-strand repairs) may withstand much greater tension than conventional two-strand sutures during early active mobilization.

However, multistrand (particularly eight-strand) repair requires complicated surgical skills; such repair is difficult. Here, we present a new eight-strand suture for flexor tendon repair that features easier passages through the tendons and fewer knots than existing approaches; it affords the necessary tensile strength to prevent both gap formation and ultimate failure.

The important aspects of flexor tendon repair are that the suture should have sufficient mechanical strength, and it should not result in a bulky configuration, which would affect tendon gliding .

Using the 8-strand repair technique and active mobilization performed by the patient is both practical and cost-saving. Intensive supervision of a hand therapist is generally not required. Notably improved outcomes have been achieved while preventing adhesions at the repair site.

ELIGIBILITY:
Inclusion Criteria

1. Adult patient
2. No fractures in the affected finger
3. Thumb is excluded
4. Duration of injury less than 2 weeks

Exclusion Criteria:

-

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
range of motion | Six month post operative
  ROM using Strickland criteria by finger goniometer

SECONDARY OUTCOMES:
Hand function | 6 month post-operative
  Hand function using DASH score
Complications | 6 month post-operative
  As rupture , adhesion

REFERENCES:
- [Background] 1.Rigo IZ, Røkkum M. Predictors of outcome after primary flexor tendon repair in zone 1, 2 and 3. J Hand Surg Eur. 2016;41:793-801. https://doi.org/10.1177/1753193416657758. Article CAS Google Scholar 2.Dy CJ, Hernandez-Soria A, Ma Y, Roberts TR, Daluiski A. Complications after flexor tendon repair: a systematic review and meta-analysis. J Hand Surg Am. 2012;37:543-551.e1. https://doi.org/10.1016/j.jhsa.2011.11.006. Article PubMed Google Scholar 3.Ishak A, Rajangam A, Khajuria A. The evidence-base for the management of flexor tendon injuries of the hand: review. Ann Med Surg. 2019;48:1-6. https://doi.org/10.1016/j.amsu.2019.10.006. Article CAS Google Scholar 4.Dy CJ, Lyman S, Schreiber JJ, Do HT, Daluiski A. The epidemiology of reoperation after flexor pulley reconstruction. J Hand Surg Am. 2013. https://doi.org/10.1016/j.jhsa.2013.05.015. Article PubMed PubMed Central Google Scholar 5.Dy CJ, Daluiski A. Update on zone II flexor tendon injuries. J Am Acad Orthop Surg. 2014. https://doi.org/10.5435/JAAOS-22-12-791. 6. Silfverskiöld K L, May E J. Flexor tendon repair in zone II with a new suture technique and an early mobilization program combining passive and active flexion. J Hand Surg Am. 1994;19(01):53-60. [PubMed] [Google Scholar] 7. Moriya K, Yoshizu T, Maki Y, Tsubokawa N, Narisawa H, Endo N. Clinical outcomes of early active mobilization following flexor tendon repair using the six-strand technique: short- and long-term evaluations. J Hand Surg Eur Vol. 2015;40(03):250-258. [PubMed] [Google Scholar] 8. Tang J B, Zhou X, Pan Z J, Qing J, Gong K T, Chen J. Strong digital flexor tendon repair, extension-flexion test, and early active flexion: experience in 300 tendons. Hand Clin. 2017;33(03):455-463. [PubMed] [Google Scholar] 9. Sandow M J, McMahon M M. Single-cross grasp six-strand repair for acute flexor tenorrhaphy: modified Savage technique. Atlas Hand Clin. 1996;1(01):41-64. [Google Scholar] 10. Yoshizu T.Immediate mobilization following flexor tendon repair(in Japanese)J Musculoskelet Syst 1996908881-890. [Google Scholar] 11. Croog A, Goldstein R, Nasser P, et al. Comparative biomechanic performances of locked cruciate four-strand flexor tendon repairs in an ex vivo porcine model. J Hand Surg Am. 2007;32:225-232. [PubMed] [Google Scholar] 12. Jordan MC, Schmitt V, Jansen H, et al. Biomechanical analysis of the modified Kessler, Lahey, Adelaide, and Becker sutures for flexor tendon repair. J Hand Surg Am. 2015;40:1812-1817. [PubMed] [Google Scholar] 13. Tarek Abdalla El-Gammal https://orcid.org/0000-0002-8434-3523 tarek.elgammal@aun.edu.eg, Mohamed Mostafa Kotb, […], and Mina Micheal Anwar+2View all authors and affiliations OnlineFirst: Outcome of Flexor Tendon Repair Using Eight-Strand Core Stitch Without Postoperative Finger Splinting, https://doi.org/10.1177/15589447231220686